CLINICAL TRIAL: NCT02781805
Title: Pilot Clinical Trial of Short-Term Bisphosphonate Administration as Chemoprevention for Breast Cancer Via Engagement of γδ T Cells
Brief Title: Pilot Study of Bisphosphonates for Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW13060; 2016-0322 (Other: Institutional Review Board); A539997 (Other: UW Madison); SMPH\VOLUNTEER STAFF\SURGERY (Other: UW Madison); NCI-2016-00786 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alendronate (Experimental): Subjects will take the study drug alendronate, a nitrogenous bisphosponate, for approximately one to three weeks before their breast surgery.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — 10 mg (1 tablet) once daily for 1-3 weeks before breast surgery; drug will be discontinued the day before surgery.
  Other Names: Fosamax; Binosto

SUMMARY:
The goal of this study is to mechanistically define the potential anticancer activities of the osteoporosis bisphosphonate (BP) drug alendronate, and extend the analysis to learn novel information about the impact of BP on gamma delta (γδ) T cells in breast tissues as well as epithelial breast cell differentiation of high-risk women. To this end, we have designed a BP "window trial" to examine the effect of 1 - 3 weeks administration of alendronate on women at high-risk for breast cancer, at the level of immunosurveillance and mammary epithelial cell differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for risk reduction mastectomy (eg. BRCA or other high-risk gene mutations, strong family history of breast cancer, prior or current LCIS, ADH, ALH and DCIS undergoing bilateral mastectomy or prophylactic contralateral mastectomy), oe patients at high-risk for breast cancer (eg. BRCA or other high-risk gene mutations, strong family history of breast cancer, prior or current LCIS, ADH, ALH and DCIS) who are not planning for immediate risk reduction mastectomy and are undergoing routine follow-up.
* Patients who are premenopausal defined as an individual with at least six menstrual cycles in the past year, women with hysterectomy with intact functioning ovaries who are not having menstrual cycles need to be 45 years of age and under.
* Patients must be 18 years of age or older
* The effects of Alendronate on the developing fetus are unknown. For this reason, sexually active heterosexual women must agree to use an effective form of birth control for the duration of study participation. Women who are NOT having 1) a hysterectomy, 2) fallopian tubes removed and/or 3) ovaries removed at the time of their breast surgery will also be required to use an effective form of birth control for 56 days following the last dose of study medication. In addition to, premenopausal women who are undergoing routine follow up and are not having surgery will be required to use an effective form of birth control for 56 days following the last dose of study medication. One of the following methods of birth control must be used by sexually active women of childbearing potential:

  * Oral contraceptive pill in continuous use for >90 days prior to study entry
  * Vaginal ring in continuous use for >90 days prior to study entry
  * Skin patch in continuous use for >90 days prior to study entry
  * Injection in continuous use prior to study entry
  * IUD
  * Diaphragm, cervical cap, or cervical shield with spermicide
  * Contraceptive sponge
  * Condom (male or female type) plus spermicide
  * Male partner who has had a vasectomy
* Women who are abstinent from heterosexual encounters for the duration of the study participation and for the 56 days following the last dose of study medication will not be required to uses birth control.
* Women with hysterectomy with intact functioning ovaries, women with Fallopian tubes cut, tied, or sealed, and women with a sterilization implant (e.g. Adiana, Essure) placed >3 months prior to beginning the study drug are not considered to be able to bear children and therefore are eligible to participate without the use of concurrent birth control.
* Females of child-bearing potential must have a negative pregnancy test within the current menstrual cycle and within 7 days before starting drug.
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* Participants must have the ability to understand, and the willingness to sign, a written informed consent form

Exclusion Criteria:

* Patients with a previous diagnosis of invasive breast cancer
* Patients who are post-menopausal (defined as 12 consecutive months without a menstrual period).
* Patients with an implant in the sampled breast
* Pregnant or lactating women are excluded from this study. Breastfeeding must be discontinued for the duration of study participation and for 8 weeks after the last dose of the study agent
* Patients for whom English is not their native language
* Patients with current or previous bisphosphonate therapy
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition of alendronate and other bisphosphonates.
* Patients with esophageal dysmotility
* Patients unable to sit up or stay up for 30 minutes after taking oral dose
* Patients who have taken non-steroidal anti-inflammatory drugs (NSAIDs) in the past two weeks
* Patients who have received chemotherapy for a malignancy in the past 5 years
* Patients who are treated for a medical condition (such as ulcerative colitis) with chronic steroids within the last 2 years
* Patients with calculated creatinine clearance (Cockroft-Gault) less than 35 mL/min
* Patients with a history of hypocalcemia
* Bilateral DCIS, LCIS, ADH or ALH

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Percentage change of γδ T cell in CNB | 1-3 weeks
  γδ T cell infiltration and activation as defined by the presence and increase in percentage of γδ T cells in the CNB sample following study agent (alendronate) administration. The effect of alendronate will be assessed using a one-tailed one-sample paired t-test or Wilcoxon signed rank test at a significance level of 0.10.

SECONDARY OUTCOMES:
Percentage change of mammary epithelial basal cells in the CNB samples after alendronate administration | 1-3 weeks
  The effect of alendronate will be assessed using a one-tailed one-sample paired t-test or Wilcoxon signed rank test at a significance level of 0.10.
Percentage change of mammary luminal cells in the CNB samples after alendronate administration | 1-3 weeks
  The effect of alendronate will be assessed using a one-tailed one-sample paired t-test or Wilcoxon signed rank test at a significance level of 0.10.

OTHER OUTCOMES:
Percentage change of γδ T cells in the blood | 1-3 weeks
  The effect of alendronate will be assessed using a one-tailed one-sample paired t-test or Wilcoxon signed rank test at a significance level of 0.10.
Ratio of percent of luminal cells to percent of basal cells in CNB | 1-3 weeks
  The effect of alendronate will be assessed using a one-tailed one-sample paired t-test or Wilcoxon signed rank test at a significance level of 0.10.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Wilke, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/